CLINICAL TRIAL: NCT05843851
Title: Scientific Basis for a Newborn Screening for Cystinosis and Primary Hyperoxaluria
Brief Title: Genetic Newborn Screening for Cystinosis and Primary Hyperoxaluria
Acronym: GENESIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cystinose Stiftung (Other)
Collaborators: Screening Laboratory Hannover (Unknown); Pediatry Kastanienhof Koeln (Unknown); Medical Genetics Mainz (Unknown); University Hospital Cologne (Unknown)
Responsible Party: Principal Investigator, Katharina Hohenfellner,MD, Head of Pediatric Nephrology, Cystinose Stiftung
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 1801-GEN-9852
Record Dates: First submitted 2023-04-11; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Cystinosis; Primary Hyperoxaluria
Keywords: Molecular based newborn screening; Cystinosis; Primary Hyperoxaluria
MeSH Terms: conditions — Cystinosis; Hyperoxaluria, Primary | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Intervention Model Description: All newborns whose parents have agreed to participate in the pilot project will be tested for two mutations in the CTNS gene and one mutation in the PH1 gene and PH 3.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tested newborns (Experimental): Tested for two mutations in the CTNS gene and one mutation in the PH1 gene and PH 3.
  Interventions: Diagnostic Test: Diagnostic test

INTERVENTIONS:
Diagnostic Test: Diagnostic test — Test for two mutations in the CTNS gene and one mutation in the PH1 gene and PH 3.

SUMMARY:
In Germany parents of newborns are offered newborn screening (NBS) for 17 congenital diseases as a standard benefit of statutory health insurance. NBS in Germany is voluntary. Cystinosis and hyperoxaluria are very rare diseases. They are inherited autosomal-recessively. Neither disease can be detected by the methods established in routine NBS. However, common genetic mutations are known for both diseases.

The aim of the study is to provide a scientific basis for molecular genetic NBS for cystinosis and primary hyperoxaluria (PH). Specifically, the study will investigate whether the inclusion of these diseases into general NBS should be recommended. By observing the identified infants in comparison to patients symptomatically diagnosed outside of the pilot project, it will be determined whether and to what extent early diagnosis and therapy lead to a more favorable prognosis.

The screening laboratory Hannover, Germany is involved in the project. Hospitals that send their dry blood spot cards for routine NBS to Hannover are offered participation in the project.

Parents who want to participate receive an additional information sheet. A parent and the attending physician sign the information sheet as documentation of informed consent, which allows data transfer and patient referral to a specialist in case of a positive result. Molecular genetic screening in the pilot project is performed from the same dry blood spot card used for routine NBS.

In both diseases, testing is performed for 2 known mutations: In cystinosis for the 2 mutations most common in Germany, and in PH for the most common mutation in infantile hyperoxaluria (PH1) and in Europe (PH3).

Normal findings are not communicated to the parents, which may contact the laboratory to ask for them. Parents of newborns with two mutations in the cystinosis gene are immediately informed about the disease by a physician. Further diagnostics to confirm the disease are organized close to home.

In contrast, parents of newborns with only one mutation in one of the two hyperoxaluria genes are informed. They are asked to send spot urines of the newborn to the hyperoxaluria center. Only if these are abnormal, further evaluation will be performed.

The study started on 15.03.2022. The aim is to screen 200,000 newborns until 2025. If the benefit of early diagnosis and therapy can be shown, an application for inclusion of a NBS for these two diseases in the routine NBS program will be submitted to the German government.

DETAILED DESCRIPTION:
Background and aims. Population-based newborn screening (NBS) is an important public health program that has vastly improved the course of several diseases through early detection. The selection of screened disorders generally follows the 10 principles outlined by Wilson and Jungner. In Germany, NBS has been a voluntary National Health Service program since 1969 which currently covers 17 disorders. Current NBS methods, which employ tandem mass-spectrometric analysis of newborn dried blood spots, cannot detect many potentially treatable genetic conditions. At the same time, molecular-based NBS is increasingly feasible because DNA can be extracted from a dried blood spot, next generation sequencing has become economical, and molecular diagnostics have greater reliability and increased validity as genetic databases become more refined and comprehensive. Nephropathic cystinosis and hyperoxaluria (PH) are eligible for molecular-based NBS because effective therapies are available.

In a first pilot project, the scientific basis for NBS for cystinosis could already be established. The aim of this study is to demonstrate the transferability of genetic NBS for Cystinosis to other laboratories and to lay the scientific basis for screening for PH.

Specifically, the study will investigate whether the inclusion of these diseases into general NBS should be recommended. By observing the identified infants in comparison to patients symptomatically diagnosed outside of the pilot project, it will be determined whether and to what extent early diagnosis and therapy lead to a more favorable prognosis.

Cystinosis Nephropathic cystinosis, due to impaired transport of cystine out of lysosomes, occurs with an incidence of 1 in 100-200,000 live births. It is characterized by renal Fanconi syndrome in the first year of life and glomerular dysfunction progression to end-stage kidney disease by approximately 10 years of age. Treatment with oral cysteamine therapy helps preserve glomerular function, but affected individuals eventually require kidney replacement therapy Cysteamine treatment generally begins at the time of diagnosis in the second year of life, but some glomerular and tubular damage has already occurred by then. This situation could be ameliorated by diagnosing patients shortly after birth, employing molecular genetics-based newborn screening. Standard mass spectrometry-based methods for newborn screening cannot detect the increased cystine content of cystinosis leukocytes.

For cystinosis screening, the first tier involved multiplex PCR to detect two of the three most common CTNS mutations in Germany. Heterozygous samples will be submitted to amplicon-based next-generation sequencing for 175 pathogenic CTNS mutations (Labor Limbach, Mainz). A detection rate of 96.5% is predicted using this approach.

Primary Hyperoxaluria Three different defaults in the glyoxylate metabolism lead to PH. The severe type PH1 is the most common variant (1-3 out of 106 patients). Population-based studies estimate a prevalence of 1:58,000. The estimated number of unreported cases is high. The deposit of calcium oxalate crystals in the kidneys triggers a chronic inflammation which results in terminal renal failure. Decreased oxalate excretion in the urine leads to high oxalate concentrations in the plasma and subsequently deposits of calcium oxalate in the organs and tissue (systemic oxalosis). The clinical course is highly variable. Examples of infantile oxalosis with early renal function loss up to a-/oligosymptomatic patients in adulthood are described.

Clinically, PH2 is calmer, but about 50% of patients develop end-stage renal failure.

PH3 used to be considered a mild variant, but it is known today that PH3 patients can also develop kidney stones in childhood and develop terminal renal failure with a systemic oxalosis.

The PH registry of OxalEurope (European hyperoxaluria consortium) currently lists 1137 genetically diagnosed patients, comprising 81.9% with PH1, 9.8% with PH2 and 8.4% with PH3. In the molecular genetic evaluation of the German registry, the results are: 74.1% PH1, 7.9% PH2 and 17% PH3.

So far, primary hyperoxaluria has been diagnosed according to clinical findings through urine analysis (or plasma test in case of terminal renal failure). Therefore, the diagnosis is usually made once patients have already developed terminal renal failure. But existing medications (Vitamin B6) or the new RNAi medications (Lumasiran, Nedosiran) can prevent renal failure and are making the disease treatable. The purpose of this pilot project is to identify the most common mutations in the AGXT gene and in the HOGA1 gene.

Workflow Study population Hospitals in Germany are free to choose between 11 certified laboratories for NBS. In this project, the Screening-Laboratory Hannover informs its senders about the possibility to extend the routinely established NBS by the genetic screening for cystinosis and PH.

The study population includes newborns whose parents wish to participate in the pilot project and have provided written informed consent.

Parent information and consent Before screening is performed, the newborn's parents are comprehensively informed about the possibility of screening for the various diseases by the physician responsible for NBS (gynecologist, pediatrician). An additional information and consent sheet for cystinosis and PH screening is inserted into the information brochure already available for regular NBS. Consent must be documented with the signature of at least one parent and the signature of the informing physician on the consent form. The consent form for the pilot project also includes consent for the transfer of contact data and findings to a specialized center in the event of an abnormal screening result. The laboratory must receive the consent form for the project prior to analysis. Results that turn out normal are reported to the responsible submitting physician according to the NBS guidelines for children. The sender must check whether there is a result for each blood sample taken for screening (result return control).

In case of a positive result, the laboratory must first inform the sender and clarify whether the child is still hospitalized. In that case, the sender obtains the initial information from the parents and notifies an expert for the respective diagnosis (Cystinosis: Priv.-Doz. Dr. med.

K. Hohenfellner, Rosenheim; Hyperoxaluria: Prof. Dr. med. B. Hoppe, Bonn). If the child has already been discharged from hospital, the laboratory will contact the relevant expert directly which is covered by the informed consent.

Sampling The molecular genetic screening is performed using the same dried blood spot card as the routine NBS.

In general, for all invalid results (i.e., if the control reaction fails) as well as all abnormal results (Cystinosis: homozygous or heterozygous for the 57-kb deletion and /or c.18_21delGACT, p.T7Ffs*7 ; PH1, c.508G>A, PH3, C700+5G>T, homozygous and/or heterozygous) the test will be internally repeated for confirmation using the existing blood sample.

Measurements and methods A real-time quadruplex PCR is performed for the four mutations described above. Cystinosis: Detection is carried out by detection of the binding or by melting analysis of fluorescence-labeled probes. In samples with a positive result due to heterozygosity mutations, the exons of the cystinosin gene (CTNS) are sequenced using next generation sequencing (NBS) in an amplicon-based method. This ensures that only the desired exons and no other DNA areas are examined. DNA already extracted for real-time multiplex PCR can be used for NBS. With NEBNext Direct Genotyping Solution all analyzable areas of CTNS gene are covered (partial overlapping), which preserve a completely sequence information of all exons and specific introns. Therefore, the DNA will be enzymatically fragmented and then ligated with illuminable adaptors. The adaptors contain individual indices. Afterwards the biotin beads will be used for the target enrichment. They will be augmented with streptavidin beads. Afterwards off-target sequences will be removed, and the libraries will be amplified by PCR. The actual sequencing is carried out using a device from Illumina (MiniSeq). The sequences are evaluated using a software that performs an automatic comparison with a reference sequence, thereby detecting mutations.

PH: The detection will be done through heat analysis with fluorescent tagged leads. In case of positive results (also due to heterozygotic constellations) a clarification is planned in collaboration with the German hyperoxaluria center. Therefore, spot urine will be tested for oxalate and further parameters in the glyoxylate metabolism.

Examination results Cystinosis: If the most frequent mutations of CTNS are detected as homozygous or compound heterozygous mutations, the cystinosis screening is considered positive. Using next-generation sequencing, an additional 175 mutations recorded in the literature will be detected. In all other cases, even those involving heterozygous status, cystinosis screening is normal.

PH: The hyperoxaluria screening is positive, if PH1 (AGXT-Gen:c508G>A) and/or PH3 (HOGA-gene: c.700+5G>T) is homozygote detected. In heterozygote genetic carrier with positive screening, a subsequent urine test performed in the Wisplinghoff laboratory in Cologne (Köln) will clarify the finding.

Detection rate, false positive and false negative results An overall detection rate of above 95% is assumed for both diseases. False negative screening results are unlikely.

For cystinosis, false negative results due to previously unknown rare mutations or patients carrying neither of the two most frequent mutations are possible.

False positive screening results are also very unlikely. With cystinosis, a heterozygous sample due to "allelic dropout" (PCR failure of an allele due to mutations in the primer binding region) may incorrectly appear homozygous.

In PH, the disease is not excluded in case of heterozygous mutation, further diagnostics is necessary and planned.

In case of corresponding symptoms, cystinosis or PH must be included in the differential diagnosis, which usually takes place in one of the few treatment centers. Such cases can only be documented in the course of time via feedback of the attending centers can be documented.

Confirmation of the diagnosis Cystinosis: In patients with either a homozygous or compound heterozygous mutation in the CTNS-gene, the diagnosis will be confirmed by determining the intraleukocytic cystine level from 2,3 ml EDTA blood. This sample will be sent to the metabolic laboratory in Heidelberg within the first 14 days of life.

PH: In homozygous carriers of the mutations in the PH1 or PH3 genes, a control examination of spot urine or of plasma will follow, which will be carried out in the German hyperoxaluria Centre.

The results of the verification tests will be transferred to the screening laboratory for quality control.

Caring for affected children Cystinosis: Children with positive cystinosis screening results and their parents are referred to the nearest center for metabolic diseases. Therapy with cysteamine can be started immediately after confirmation of the diagnosis. Parents are informed about the possibility of an interdisciplinary cystinosis consultation in Rosenheim.

PH: Children with a positive screening result will be primarily referred to the German hyperoxaluria center in Bonn.

Further treatment of these patients is performed at the nearest hospital of their choice.

Project size For financial reasons, the project is limited to 200,000 samples, with the possibility of expansion.

ELIGIBILITY:
Inclusion Criteria:

* Newborns participating at the NGS with parent's consent to participate in this screening project

Exclusion Criteria:

* Newborns without parent's consent to participate in this screening project.

Ages: 32 Hours to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200000 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Newborns with confirmed diagnosis of Cystinosis | 12 months
  Newborns identified with 57-kb CTNS mutation homozygous, compound heterozygous, with c.18_21delGACT p.T7Ffs*7 homozygous or compound heterozygous and elevated white blood cell cystine level.
Number of newborns with heterozygous mutations | 12 months
  Newborns identified with heterozygous CTNS mutations of 57-kb CTNS and heterozygous c.18_21delGACT p.T7Ffs*7 mutations
Patients with PH1 and PH3 | 12 months
  Newborns identified with heterozygous PH1 c.508G>A and PH3, C700+5G>T and further positive evaluation of urine and genetic analysis.

SECONDARY OUTCOMES:
Newborns identified with heterozygous PH1 c.508G>A and PH3, C700+5G>T | 12 months
  Results of urine analysis of patients with heterozygous PH1 c.508G>A and PH3, C700+5G>T

OTHER OUTCOMES:
Both diseases | time interval until start of treatment
  For both diseases the time interval will be evaluated from the time of identification in screening to the introduction of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Sonja Froschauer, Study Director — Cystinosis Foundation (Cystinose Stiftung); Katharina Hohenfellner, Study Chair — Ro Med Clinics Rosenheim
Locations (1):
- Screening Laboratory Hanover, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No
Due to foundation legal requirements, no further information can be shared.

REFERENCES:
- [Background] Hohenfellner K, Bergmann C, Fleige T, Janzen N, Burggraf S, Olgemoller B, Gahl WA, Czibere L, Froschauer S, Roschinger W, Vill K, Harms E, Nennstiel U. Molecular based newborn screening in Germany: Follow-up for cystinosis. Mol Genet Metab Rep. 2019 Sep 18;21:100514. doi: 10.1016/j.ymgmr.2019.100514. eCollection 2019 Dec. PMID 31641587
- [Background] Fleige T, Burggraf S, Czibere L, Haring J, Gluck B, Keitel LM, Landt O, Harms E, Hohenfellner K, Durner J, Roschinger W, Becker M. Next generation sequencing as second-tier test in high-throughput newborn screening for nephropathic cystinosis. Eur J Hum Genet. 2020 Feb;28(2):193-201. doi: 10.1038/s41431-019-0521-3. Epub 2019 Sep 30. PMID 31570786
- [Background] Niessl C, Boulesteix AL, Oh J, Palm K, Schlingmann P, Wygoda S, Haffner D, Wuhl E, Tonshoff B, Buescher A, Billing H, Hoppe B, Zirngibl M, Kettwig M, Moeller K, Acham-Roschitz B, Arbeiter K, Bald M, Benz M, Galiano M, John-Kroegel U, Klaus G, Marx-Berger D, Moser K, Mueller D, Patzer L, Pohl M, Seitz B, Treikauskas U, von Vigier RO, Gahl WA, Hohenfellner K. Relationship between age at initiation of cysteamine treatment, adherence with therapy, and glomerular kidney function in infantile nephropathic cystinosis. Mol Genet Metab. 2022 Aug;136(4):268-273. doi: 10.1016/j.ymgme.2022.06.010. Epub 2022 Jul 2. PMID 35835062
- [Background] Hohenfellner K, Niessl C, Haffner D, Oh J, Okorn C, Palm K, Schlingmann KP, Wygoda S, Gahl WA. Beneficial effects of starting oral cysteamine treatment in the first 2 months of life on glomerular and tubular kidney function in infantile nephropathic cystinosis. Mol Genet Metab. 2022 Aug;136(4):282-288. doi: 10.1016/j.ymgme.2022.06.009. Epub 2022 Jul 1. PMID 35843134
- [Background] Hopp K, Cogal AG, Bergstralh EJ, Seide BM, Olson JB, Meek AM, Lieske JC, Milliner DS, Harris PC; Rare Kidney Stone Consortium. Phenotype-Genotype Correlations and Estimated Carrier Frequencies of Primary Hyperoxaluria. J Am Soc Nephrol. 2015 Oct;26(10):2559-70. doi: 10.1681/ASN.2014070698. Epub 2015 Feb 2. PMID 25644115
- [Background] Garrelfs SF, Rumsby G, Peters-Sengers H, Erger F, Groothoff JW, Beck BB, Oosterveld MJS, Pelle A, Neuhaus T, Adams B, Cochat P, Salido E, Lipkin GW, Hoppe B, Hulton SA; OxalEurope Consortium. Patients with primary hyperoxaluria type 2 have significant morbidity and require careful follow-up. Kidney Int. 2019 Dec;96(6):1389-1399. doi: 10.1016/j.kint.2019.08.018. Epub 2019 Sep 3. PMID 31685312
- [Background] Hoyer-Kuhn H, Kohbrok S, Volland R, Franklin J, Hero B, Beck BB, Hoppe B. Vitamin B6 in primary hyperoxaluria I: first prospective trial after 40 years of practice. Clin J Am Soc Nephrol. 2014 Mar;9(3):468-77. doi: 10.2215/CJN.06820613. Epub 2014 Jan 2. PMID 24385516
- [Background] Hoppe B, Koch A, Cochat P, Garrelfs SF, Baum MA, Groothoff JW, Lipkin G, Coenen M, Schalk G, Amrite A, McDougall D, Barrios K, Langman CB. Safety, pharmacodynamics, and exposure-response modeling results from a first-in-human phase 1 study of nedosiran (PHYOX1) in primary hyperoxaluria. Kidney Int. 2022 Mar;101(3):626-634. doi: 10.1016/j.kint.2021.08.015. Epub 2021 Sep 2. PMID 34481803
- [Background] Hoppe B, Martin-Higueras C. Improving Treatment Options for Primary Hyperoxaluria. Drugs. 2022 Jul;82(10):1077-1094. doi: 10.1007/s40265-022-01735-x. Epub 2022 Jul 2. PMID 35779234
- [Background] Elmonem MA, Veys KR, Soliman NA, van Dyck M, van den Heuvel LP, Levtchenko E. Cystinosis: a review. Orphanet J Rare Dis. 2016 Apr 22;11:47. doi: 10.1186/s13023-016-0426-y. PMID 27102039